CLINICAL TRIAL: NCT07273279
Title: Associations of ADH1B and ALDH Family Gene Polymorphisms With Lung Cancer Risk and Its Subtypes: Results From the Oncoarray Project of the International Lung Cancer Consortium
Brief Title: ADH1B and ALDH Gene Variants and Lung Cancer Risk
Acronym: ALDH
Status: Not yet recruiting | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Tzu Yu Pan, Postdoctoral Researcher, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUHIRB-E(I)-20250145; 113-2314-B-037 -070 -MY3 (Other: National Science and Technology Council (Taiwan))
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Condition/Disease; Lung Cancer (Diagnosis); Lung Adenocarcinoma
Keywords: ALDH2; ADH1B; Lung cancer
MeSH Terms: conditions — Disease; Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer in never-smokers is increasingly recognized as a disease influenced by genetic susceptibility. Aldehyde-metabolizing enzymes, including the ALDH gene family and ADH1B, play key roles in detoxifying reactive aldehydes that can damage DNA and promote oxidative stress. In this study, we will examine whether ten selected genetic variants, nine single nucleotide polymorphisms (SNPs) across five ALDH family genes and one variant in ADH1B are associated with the risk of lung cancer and its major subtypes. Limited epidemiological evidence is currently available on the association between these aldehyde-metabolizing gene variants and lung cancer. This research aims to clarify their potential contribution to the development of lung cancer, particularly among never-smokers.

DETAILED DESCRIPTION:
This case-control study aims to investigate the association of ten genetic variants-nine SNPs across five ALDH family genes and one SNP in ADH1B (rs1229984)-with the risk of lung cancer and its major subtypes. The primary hypothesis is that the ALDH2 rs671 variant is associated with the risk of lung cancer and its major subtypes. The secondary hypothesis is that other ALDH variants-including rs2228093 and rs2073478 in ALDH1B1, rs1127717 and rs2276724 in ALDH1L1, rs3741172, rs17856219, and rs77341916 in ALDH3B2, and rs3765310 in ALDH5A1-are also associated with lung cancer risk. Demographic and lifestyle covariates such as age, gender, ethnicity, smoking status, alcohol consumption, educational level, and case-control status will be incorporated into the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Incident lung cancer cases confirmed by pathology and healthy adult over age of 18 years.

Exclusion Criteria:

* Individuals with incomplete data will not be included as study participants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung cancer status determined by pathology-confirmed diagnosis at the time of case identification
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Lung cancer status (case vs control) | Not applicable (baseline status)
  Lung cancer status determined by pathology-confirmed diagnosis at the time of case identification

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because data use agreements restrict redistribution of participant-level data.